CLINICAL TRIAL: NCT06212479
Title: A Multi-Site Prospective, Single-Arm, Observational Study On The Accuracy Of Whole Body Magnetic Resonance Imaging (Wb-Mri) Screening To Predict Clinically Significant Diagnoses In General Population Subjects Interested In Proactive And Advanced General Preventive Healthcare.
Brief Title: An Observational Study On TheAccuracy Of Whole-Body Magnetic Resonance Imaging (Wb-Mri) ScreeningTo Predict Clinically Significant Diagnoses In General Population Subjects Interested In Proactive And Advanced General Preventive Healthcare.
Acronym: Hercules
Status: Recruiting | Type: Observational
Sponsor: Hercules (Industry)
Collaborators: Prenuvo Inc (Unknown)
Responsible Party: Sponsor
Other Study IDs: MA- 001
Record Dates: First submitted 2023-12-26; First posted 2024-01-18 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Cancer; Metabolic Disease; Aneurysm; Neurologic Disorder
MeSH Terms: conditions — Neoplasms; Metabolic Diseases; Aneurysm; Nervous System Diseases | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MRI Scan Arm: Whole Body MRI Scan
  Interventions: Diagnostic Test: MRI Scan

INTERVENTIONS:
Diagnostic Test: MRI Scan — Whole Body MRI Scan

SUMMARY:
This is a prospective, single-arm, observational study capturing data from whole-body magnetic resonance imagining (WB-MRI) from up to 100,000 male and female subjects 18 years of age or older recruited at multiple clinical sites within the United States. Study subjects must meet a set of inclusion and exclusion criteria. Potential subjects arriving at the study sites will be evaluated for enrollment. It is the Principal Investigator's (PI) responsibility to enroll only subjects who satisfy the inclusion/exclusion criteria. Recruitment can occur by subject presentation at the sites for elective standard screening, word-of-mouth, flyers, healthcare professional (HCP) referrals, advertisement online, or any other means, subject to approval by the associated institutional review board (IRB) or ethics committee (EC) when applicable.

ELIGIBILITY:
Inclusion Criteria:

* Each subject MUST:

  * Be>=18 years of age at the time of enrollment.
  * Be able to read and understand provided procedural information for the study;
  * Be able and willing to follow all study procedures including proper breathing and body movement minimization while within the WB-MRI system;
  * Be willing and able to provide required clinical, demographic, medical history, and concomitant medications information;
  * Be able to provide financial payment in advance for reimbursement of the cost of the WBMRI acquisition procedure and interpretation;
  * Complete all required consent procedures.

Exclusion Criteria:

* Harbor within their bodies contraindicated medical devices including, but not limited to, implanted pacemakers, intracranial aneurysm clips, cochlear implants, drug infusion pumps, neurostimulators, bone growth stimulators, certain intrauterine contraceptive devices, non- MRI safe metals, etc.;

  * Self-certify that they are pregnant;
  * Be seeking to undergo WB-MRI as a subject in this study in lieu of other covered dedicated diagnostic imaging evaluations when such covered procedures represent more appropriate or standard-of-care procedures by context-specific clinical indication;
  * Be an employee of the study site or the sponsor;
  * Have a medical condition or serious intercurrent illness, or other circumstance that, in the Investigator's judgment, could jeopardize the candidate's safety as a study subject, or that could interfere with study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All the patients above 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2034-01 (Estimated); Study Completion 2037-01 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint and 5-point scale of CSD (Clinically Significant Disease) of CSD diagnosed post-baseline in general population subjects. | Up to 10 Years
  Clinically significant disease represents the primary output of WB-MRI image analysis, and thus, the primary endpoint for this study. This outcome will be expressed as a 5-point scale similar to the standard Likert scale used in clinical studies. Higher the number higher the risk of clinically significant finding.

SECONDARY OUTCOMES:
Secondary Endpoint of ONCO-RADS Score (Oncological relevant findings reporting and data system) diagnosed in the follow-up period, including but not limited to, types of cancers, aneurysms, metabolic disorders, neurologic disorders, renal function, etc | Up to 10 Years
  Additionally, for the purposes of more specifically distinguishing CSD's of oncological-concern, following the ONCO-RADS7 guidelines for cancer screening utilizing WB-MRI, an additional ONCO-RADS score tag ("ONCO") will be attached to each CSD to reflect oncologic-specific risk according to the screening WB-MRI criteria. Higher the number worse the risk of having Cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Perry Kaneriya, MD, MBA, Principal Investigator — Hercules
Locations (1):
- Hercules Research Center, Watertown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided